CLINICAL TRIAL: NCT00289432
Title: Effects of Group Intervention on Anxiety, Depression and Quality of Life Among Women Operated for Breast Cancer. A Randomized, Prospective Study.
Brief Title: Hospital Based Group Intervention for Breast Cancer Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Principal Investigator, Inger Schou Bredal, Associate Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: INCAM
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer; Anxiety; Depression; Quality of Life; Coping
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Behavioral: Psychoeducative intervention
  Interventions: Behavioral: Psychoeducative
- 2 (Active Comparator): The Hospitals standard follow-up support group
  Interventions: Other: Support group

INTERVENTIONS:
Behavioral: Psychoeducative — The experimental group consists of five weekly 2-hours sessions, focusing on coping with diagnosis and treatment
  Other Names: Intervention group
  Arms: 1
Other: Support group — Standard Hospital follow-up support group
  Other Names: Standard group
  Arms: 2

SUMMARY:
INCAM-study is a multicenter, prospective, randomized controlled trial. The aim of the study is to test the effectiveness of psychoeducative intervention when offered in hospital setting as a component of routine breast cancer care. The hypotheses are; - that breast cancer patients participating in psychoeducative interventions focusing on coping will experience better health-related quality of life than those who participate in the hospital standardised psychoeducative intervention. - that coping styles are associated with the immune system.

DETAILED DESCRIPTION:
Women operated for breast cancer often experience psychosocial problems for several years. Although, meta-analyses have clearly demonstrated that the efficacy of psychosocial support groups, little is known about the effectiveness of this intervention when offered in the hospital setting as a component of routine breast cancer care.

A few studies have found that psychological intervention reduce emotional distress and enhance immune responses,but if there is an association between coping styles and immune system is not clear.

440 breast cancer patients at two Hospital will be randomized into the study. Both Hospital have standardised psychoeducative interventions as a component of routine breast cancer care. Both Hospital will have two groups, the standardised groups and the experimental groups. Participants will answer the same standardised questionnaires before surgery,2,6,12 months and 3 and 5 years after the interventions. Blood sample will be drawn at all assessments. The questionnaires are the Hospital Anxiety and Depression Scale, the Mini-mental Adjustment to Cancer Scale, the EORTC QLQ-BR32, the Life Orientation Test-Revised.

All groups are facilitated by two nurse specialists and follow a structured program. The standardised groups consists of three weekly 2-hours sessions and the experimental groups will consists of six weekly 2-hours session. The intervention protocol has been approved by the Norwegian Committee for medical research Ethics.

Knowledge from this study will be used to develop a manual for hospital based group interventions for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Verified breast cancer diagnosis Age 18 years or more but under 75 years -

Exclusion Criteria:

Diagnoses of metastatic breast cancer Do not read or write Norwegian Diagnoses of mental retardation, severe or untreated psychopathology, dementia Diagnoses of any immunologic condition or disease

-

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2006-04; Primary Completion 2009-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Scores on Health-related quality of life | 2, 6 12 months and at 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Inger Schou Bredal, PhD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Oslo County, Norway